CLINICAL TRIAL: NCT01427322
Title: A Randomized Study of Lapatinib With Radiation Versus Radiation Alone in Advanced Solid Tumor Cancer Patients Receiving Radiation Therapy for Metastatic Disease
Brief Title: Randomized RT +/- Lapatinib for Advanced Solid Tumor Cancer Patients Receiving Radiation Therapy for Metastatic Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13711; NCI-2011-02734 (Registry Identifier: CTRP)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Epithelial Cancer
Keywords: lapatinib; radiation therapy; metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Lapatinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lapatinib + radiation therapy (Experimental): lapatinib given orally 2-4 hours prior to first fraction of radiation
  Interventions: Drug: Lapatinib; Radiation: Radiation therapy
- No therapy prior to radiation (Active Comparator): Radiation therapy alone
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Drug: Lapatinib — given orally 2-4 hours before first fraction of radiation therapy
  Other Names: GW572016; Tykerb
  Arms: lapatinib + radiation therapy
Radiation: Radiation therapy — Standard radiation therapy

SUMMARY:
Lapatinib will prevent radiation-induced increase in Transforming Growth Factor alpha (TGFα), an important growth factor in cancer cell recovery after ionizing irradiation.

DETAILED DESCRIPTION:
Lapatinib is an orally bioavailable small molecule inhibitor of ERBB1 and ERBB2 (HER2). It is currently indicated for use in patients with HER2 over-expressing metastatic breast cancer. Serum increases in TGFα can have growth potentiating effects on distant sites of metastatic disease. Palliative irradiation paradoxically may promote distant tumor growth; blocking shedding of TGFα from irradiated tumors may prevent this effect and improve the therapeutic index of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* History of stage IV epithelial-derived cancer requiring palliative radiation. Patients with sarcoma, lymphoma, myeloma or neuroendocrin cancers are not eligible.
* Evidence of metastatic disease
* Recommendation by patient's radiation oncologist to receive palliative external beam radiation for metastases -- minimum fraction size of 3 Gy.
* Age 18 years or older
* Patients may be undergoing concurrent therapy with GNRH agonists or combined androgen blockade or anti-estrogen hormonal therapy for breast cancer, as these are standard care for advanced prostate and some breast cancers respectively.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any contraindication to lapatinib treatment.
* Prior radiation therapy within 30 days of the start of the planned course of treatment.
* Prior cytotoxic chemotherapy within 4-2 weeks of planned first dose of radiation. Persistent grade 2 or greater non-hematologic toxicity (other than neuropathy) from cytotoxic chemotherapy regardless of interval since last dose. Persistent grade 3 or greater hematologic toxicity (other than lymphopenia) reglardless of interval since last dose.
* Prior administration of an ERBB1 or ERK1/2 inhibitor within 30 days of the start of the planned course of treatment.
* Patients with a medical necessity to continue active therapy with CYP3A4 strong inhibitors or inducers. The concomitant use of strong CYP3A4 inhibitors should be avoided (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, aprepitant). Grapefruit may also increase plasma concentrations of lapatinib and should be avoided. Once the strong inhibitor or inducer is discontinued, a washout period of approximately 1 week should be allowed before the lapatinib administration. If a patient is unable to discontinue these medications, they are not eligible for enrollment.
* Concurrent administration of any other investigational agents.
* Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active hepatic or biliary disease with a Child-Pugh class of B or C, or psychiatric illness/social situations that would limit compliance with study requirements or that would interfere with accomplishing the study objectives.
* Pregnant or nursing. Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to the start of treatment. Women of childbearing potential and men must agree to use a medically accepted form of birth control for the duration of study participation. Men must agree to use a medically accepted form of birth control for 4 months following completion of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
TGFalpha | 3 years
  Blockade of the ERBB1 receptor will abrogate increases in TGFalpha in response to radiation therapy. We will compare serum changes in TGFalpha between the lapatinib and control groups for patients receiving radiotherapy for stage IV epithelial-derived cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Poklepovic, MD, Principal Investigator — Massey Cancer Center
Locations (2):
- United States (2):
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Massey Cancer Center, Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- See also: Massey Cancer Center — http://www.massey.vcu.edu/